CLINICAL TRIAL: NCT03212352
Title: Mifepristone and Misoprostol Versus Misoprostol Alone for Uterine Evacuation After Early Pregnancy Failure: a Randomized Double Blind Placebo-controlled Comparison (Triple M Trial)
Brief Title: Comparing Two Medical Treatments for Early Pregnancy Failure.
Acronym: Triple M
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Advised by DSMB based on interim-analysis, highly significant difference.
Sponsor: Radboud University Medical Center (Other)
Collaborators: Innovatiefonds Zorgverzekeraars (Other); Canisius-Wilhelmina Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 62449
Record Dates: First submitted 2017-07-02; First posted 2017-07-11 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2019-09

CONDITIONS: Early Pregnancy Failure
Keywords: miscarriage; mifepristone; misoprostol; medical treatment; patient satisfaction; abortifacient agents
MeSH Terms: conditions — Abortion, Spontaneous; Patient Satisfaction | interventions — Mifepristone; Misoprostol

STUDY DESIGN:
Intervention Model Description: Before medical treatment with misoprostol (two doses 400mcg (four hours apart), repeated after 24 hours if no tissue is lost), patients will be randomized to oral mifepristone (600mg) or oral placebo (identical in appearance).
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Misoprostol (Placebo Comparator): Before medical treatment with misoprostol (two doses 400mcg (four hours apart), repeated after 24 hours if no tissue is lost), patients receive an oral placebo.
  Interventions: Drug: Misoprostol
- Misoprostol and Mifepristone (Experimental): Before medical treatment with misoprostol (two doses 400mcg (four hours apart), repeated after 24 hours if no tissue is lost), patients receive oral mifepristone (600mg).
  Interventions: Drug: Mifepristone; Drug: Misoprostol

INTERVENTIONS:
Drug: Mifepristone — Adding 600 mg of Mifepristone to the regular treatment with Misoprostol 800 mcg.
  Other Names: Mifegyne
  Arms: Misoprostol and Mifepristone
Drug: Misoprostol — Regular treatment with Misoprostol 800 mcg.
  Other Names: Cytotec

SUMMARY:
This study aims to compare whether a combination of two drugs (Mifepristone and misoprostol) are superior compared to using only one of these drugs (Misoprostol) as medical treatment for a miscarriage. Women in whom early pregnancy failure, 6-14 weeks postmenstrual, is ultrasonographically confirmed qualify for this study.

It is expected that the combination of Mifepristone and Misoprostol is more effective in reaching complete evacuation, and therefore can prevent more invasive treatment such as curettage.

DETAILED DESCRIPTION:
This study will test the hypothesis that, in early pregnancy failure, the sequential combination of mifepristone with misoprostol is superior to the use of misoprostol alone in terms of complete evacuation of products of conception (primary outcome), patient satisfaction, complications, side effects and costs (secondary outcomes). The trial will be performed multi-centred (hospitals), prospectively, two-armed, randomized, double-blinded and placebo-controlled.

Women with ultrasonographically confirmed early pregnancy failure (6-14 weeks postmenstrual), managed expectantly for at least one week, can be included. Before medical treatment with misoprostol (two doses 400mcg (four hours apart), repeated after 24 hours if no tissue is lost), patients will be randomized to oral mifepristone (600mg) or oral placebo (identical in appearance). The investigators aim to randomize 460 women in a 1:1 ratio, stratified by centre.

After six weeks, the primary endpoint, complete or incomplete evacuation, will be determined

ELIGIBILITY:
Inclusion Criteria:

Early pregnancy failure, 6-14 weeks postmenstrual with

* a crown-rump length ≥ 6mm and no cardiac activity OR
* a crown-rump length <6mm and no fetal growth at least one week later OR
* a gestational sac with absent embryonic pole for at least one week.

  * At least one week after diagnosis OR a discrepancy of at least one week between crown-rump length and calendar gestational age
  * Intra-uterine pregnancy
  * Women aged above 16 years
  * Hemodynamic stable patient
  * No signs of infection
  * No signs of incomplete abortion
  * No contraindications for mifepristone or misoprostol

Exclusion Criteria:

* Patient does not meet inclusion criteria, discovered after randomization
* Inability to give informed consent
* Known clotting disorder or use of anticoagulants
* Known risk factors for, or presence of, a cardiovascular disease
* Language barrier

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 342 (Actual)
Dates: Start 2018-06-27 (Actual); Primary Completion 2020-01-23 (Actual); Study Completion 2020-03-16 (Actual)

PRIMARY OUTCOMES:
Complete evacuation | six weeks after initial treatment
  Whether or not complete evacuation (total endometrial thickness <15 mm) has been acquired will be assessed through ultrasonography.

SECONDARY OUTCOMES:
patient satisfaction | At baseline, day four, two and six weeks after treatment
  To assess how satisfied patient are with the treatment they underwent. Patient satisfaction with treatment will be measured using The Client Satisfaction Questionnaire (CSQ-8, digital)
complications | six weeks after treatment
  How many and which complications have occured?
side effects | six weeks after treatment
  Which side effects have patients experienced and to what degree?
costs | up to six weeks after treatment
  To evaluate which medical treatment strategy is cost-effective, volumes of health care consumed will additionally be measured prospectively alongside the clinical trial together with cost associated with productivity losses. Costs of medical interventions (direct costs) and costs resulting from productivity loss (indirect costs) will be taken into account. Resource uses will be recorded in the case report forms. Standardized unit costs will be calculated using the Dutch manual for costing in economic evaluations and standardised costs.
Overall quality of health, as experienced by the patient. | At baseline, day four, and two and six weeks after initial treatment.
  To measure the quality of the health status of the patients, a validated so-called health-related quality of life (HRQoL) instrument will be used: the Short Form 36 health survey
Overall quality of health, as experienced by the patient. | At baseline, day four, and two and six weeks after initial treatment.
  To measure the quality of the health status of the patients,a validated so-called health-related quality of life (HRQoL) instrument will be used: the EuroQol-5D.

CONTACTS AND LOCATIONS:
Overall Officials: Frank P. Vandenbussche, Prof. Dr., Study Director — Radboud University Medical Center
Locations (13):
- Netherlands (13):
  - Rijnstate, Arnhem, Gelderland
  - Radboud University Medical Centre, Nijmegen, Gelderland
  - Canisius Wilhelmina Hospital, Nijmegen, Gelderland
  - Maasstad Ziekenhuis, Rotterdam, South Holland
  - OLVG, Amsterdam
  - Amphia Hospital, Breda
  - Catharina Hospital, Eindhoven
  - Martini Hospital, Groningen
  - Zuyderland Medical Centre, Heerlen
  - St. Antonius Hospital, Nieuwegein
  - Laurentius Hosptial, Roermond
  - Haaglanden Medical Centre, The Hague
  - VieCuri Medical Centre, Venlo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Graziosi GC, Mol BW, Reuwer PJ, Drogtrop A, Bruinse HW. Misoprostol versus curettage in women with early pregnancy failure after initial expectant management: a randomized trial. Hum Reprod. 2004 Aug;19(8):1894-9. doi: 10.1093/humrep/deh344. Epub 2004 Jun 10. PMID 15192065
- [Background] You JH, Chung TK. Expectant, medical or surgical treatment for spontaneous abortion in first trimester of pregnancy: a cost analysis. Hum Reprod. 2005 Oct;20(10):2873-8. doi: 10.1093/humrep/dei163. Epub 2005 Jun 24. PMID 15979988
- [Background] Hooker AB, Lemmers M, Thurkow AL, Heymans MW, Opmeer BC, Brolmann HA, Mol BW, Huirne JA. Systematic review and meta-analysis of intrauterine adhesions after miscarriage: prevalence, risk factors and long-term reproductive outcome. Hum Reprod Update. 2014 Mar-Apr;20(2):262-78. doi: 10.1093/humupd/dmt045. Epub 2013 Sep 29. PMID 24082042
- [Background] Lemmers M, Verschoor MA, Hooker AB, Opmeer BC, Limpens J, Huirne JA, Ankum WM, Mol BW. Dilatation and curettage increases the risk of subsequent preterm birth: a systematic review and meta-analysis. Hum Reprod. 2016 Jan;31(1):34-45. doi: 10.1093/humrep/dev274. Epub 2015 Nov 2. PMID 26534897
- [Background] Soulat C, Gelly M. [Immediate complications of surgical abortion]. J Gynecol Obstet Biol Reprod (Paris). 2006 Apr;35(2):157-62. doi: 10.1016/s0368-2315(06)76389-x. French. PMID 16575361
- [Background] Niinimaki M, Jouppila P, Martikainen H, Talvensaari-Mattila A. A randomized study comparing efficacy and patient satisfaction in medical or surgical treatment of miscarriage. Fertil Steril. 2006 Aug;86(2):367-72. doi: 10.1016/j.fertnstert.2005.12.072. Epub 2006 Jun 9. PMID 16764872
- [Background] Neilson JP, Hickey M, Vazquez J. Medical treatment for early fetal death (less than 24 weeks). Cochrane Database Syst Rev. 2006 Jul 19;2006(3):CD002253. doi: 10.1002/14651858.CD002253.pub3. PMID 16855990
- [Background] van den Berg J, Gordon BBM, Snijders MPML, Vandenbussche FPHA, Coppus SFPJ. The added value of mifepristone to non-surgical treatment regimens for uterine evacuation in case of early pregnancy failure: a systematic review of the literature. Eur J Obstet Gynecol Reprod Biol. 2015 Dec;195:18-26. doi: 10.1016/j.ejogrb.2015.09.027. Epub 2015 Sep 30. PMID 26461963
- [Background] Lemmers M, Verschoor MAC, Oude Rengerink K, Naaktgeboren C, Bossuyt PM, Huirne JAF, Janssen IAH, Radder C, Klinkert ER, Langenveld J, van der Voet L, Siemens FF, Bongers MY, van Hooff MH, van der Ploeg M, Sjors FPJ, Coppus SFPJ, Ankum WM, Mol BWJ; MisoREST study group. MisoREST: Surgical versus expectant management in women with an incomplete evacuation of the uterus after misoprostol treatment for miscarriage: A cohort study. Eur J Obstet Gynecol Reprod Biol. 2017 Apr;211:83-89. doi: 10.1016/j.ejogrb.2017.01.019. Epub 2017 Jan 27. PMID 28209537
- [Background] Lemmers M, Verschoor MA, Oude Rengerink K, Naaktgeboren C, Opmeer BC, Bossuyt PM, Huirne JA, Janssen CA, Radder C, Klinkert ER, Langenveld J, Catshoek R, Van der Voet L, Siemens F, Geomini P, Van Hooff MH, Van der Ploeg JM, Coppus SF, Ankum WM, Mol BW; MisoREST study group. MisoREST: surgical versus expectant management in women with an incomplete evacuation of the uterus after misoprostol treatment for miscarriage: a randomized controlled trial. Hum Reprod. 2016 Nov;31(11):2421-2427. doi: 10.1093/humrep/dew221. Epub 2016 Sep 2. PMID 27591236
- [Background] Say L, Kulier R, Gulmezoglu M, Campana A. Medical versus surgical methods for first trimester termination of pregnancy. Cochrane Database Syst Rev. 2005 Jan 25;2002(1):CD003037. doi: 10.1002/14651858.CD003037.pub2. PMID 15674900
- [Background] Kulier R, Kapp N, Gulmezoglu AM, Hofmeyr GJ, Cheng L, Campana A. Medical methods for first trimester abortion. Cochrane Database Syst Rev. 2011 Nov 9;2011(11):CD002855. doi: 10.1002/14651858.CD002855.pub4. PMID 22071804
- [Background] Maria B, Chaneac M, Stampf F, Ulmann A. [Early pregnancy interruption using an antiprogesterone steroid: Mifepristone (RU 486)]. J Gynecol Obstet Biol Reprod (Paris). 1988;17(8):1089-94. French. PMID 3235788
- [Background] Grimes DA, Mishell DR Jr, Shoupe D, Lacarra M. Early abortion with a single dose of the antiprogestin RU-486. Am J Obstet Gynecol. 1988 Jun;158(6 Pt 1):1307-12. doi: 10.1016/0002-9378(88)90361-4. PMID 2454578
- [Background] van den Berg J, van den Bent JM, Snijders MP, de Heus R, Coppus SF, Vandenbussche FP. Sequential use of mifepristone and misoprostol in treatment of early pregnancy failure appears more effective than misoprostol alone: a retrospective study. Eur J Obstet Gynecol Reprod Biol. 2014 Dec;183:16-9. doi: 10.1016/j.ejogrb.2014.10.010. Epub 2014 Oct 14. PMID 25461345
- [Background] Stockheim D, Machtinger R, Wiser A, Dulitzky M, Soriano D, Goldenberg M, Schiff E, Seidman DS. A randomized prospective study of misoprostol or mifepristone followed by misoprostol when needed for the treatment of women with early pregnancy failure. Fertil Steril. 2006 Oct;86(4):956-60. doi: 10.1016/j.fertnstert.2006.03.032. PMID 17027362
- [Background] Wagaarachchi PT, Ashok PW, Narvekar N, Smith NC, Templeton A. Medical management of early fetal demise using a combination of mifepristone and misoprostol. Hum Reprod. 2001 Sep;16(9):1849-53. doi: 10.1093/humrep/16.9.1849. PMID 11527887
- [Background] Gronlund A, Gronlund L, Clevin L, Andersen B, Palmgren N, Lidegaard O. Management of missed abortion: comparison of medical treatment with either mifepristone + misoprostol or misoprostol alone with surgical evacuation. A multi-center trial in Copenhagen county, Denmark. Acta Obstet Gynecol Scand. 2002 Nov;81(11):1060-5. PMID 12421175
- [Background] Coughlin LB, Roberts D, Haddad NG, Long A. Medical management of first trimester miscarriage (blighted ovum and missed abortion): is it effective? J Obstet Gynaecol. 2004 Jan;24(1):69-71. doi: 10.1080/01443610310001620332. PMID 14675986
- [Background] Schreiber CA, Creinin MD, Reeves MF, Harwood BJ. Mifepristone and misoprostol for the treatment of early pregnancy failure: a pilot clinical trial. Contraception. 2006 Dec;74(6):458-62. doi: 10.1016/j.contraception.2006.07.007. Epub 2006 Sep 7. PMID 17157102
- [Background] Kollitz KM, Meyn LA, Lohr PA, Creinin MD. Mifepristone and misoprostol for early pregnancy failure: a cohort analysis. Am J Obstet Gynecol. 2011 May;204(5):386.e1-6. doi: 10.1016/j.ajog.2010.12.026. Epub 2011 Feb 8. PMID 21306697
- [Background] Torre A, Huchon C, Bussieres L, Machevin E, Camus E, Fauconnier A. Immediate versus delayed medical treatment for first-trimester miscarriage: a randomized trial. Am J Obstet Gynecol. 2012 Mar;206(3):215.e1-6. doi: 10.1016/j.ajog.2011.12.009. Epub 2011 Dec 16. PMID 22381604
- [Background] Luise C, Jermy K, May C, Costello G, Collins WP, Bourne TH. Outcome of expectant management of spontaneous first trimester miscarriage: observational study. BMJ. 2002 Apr 13;324(7342):873-5. doi: 10.1136/bmj.324.7342.873. PMID 11950733
- [Background] Rulin MC, Bornstein SG, Campbell JD. The reliability of ultrasonography in the management of spontaneous abortion, clinically thought to be complete: a prospective study. Am J Obstet Gynecol. 1993 Jan;168(1 Pt 1):12-5. doi: 10.1016/s0002-9378(12)90877-7. PMID 8420312
- [Background] Creinin MD, Harwood B, Guido RS, Fox MC, Zhang J; NICHD Management of Early Pregnancy Failure Trial. Endometrial thickness after misoprostol use for early pregnancy failure. Int J Gynaecol Obstet. 2004 Jul;86(1):22-6. doi: 10.1016/j.ijgo.2004.02.004. PMID 15207665
- [Background] Chung TK, Cheung LP, Sahota DS, Haines CJ, Chang AM. Evaluation of the accuracy of transvaginal sonography for the assessment of retained products of conception after spontaneous abortion. Gynecol Obstet Invest. 1998;45(3):190-3. doi: 10.1159/000009954. PMID 9565145
- [Background] Jauniaux E, Johns J, Burton GJ. The role of ultrasound imaging in diagnosing and investigating early pregnancy failure. Ultrasound Obstet Gynecol. 2005 Jun;25(6):613-24. doi: 10.1002/uog.1892. PMID 15861413
- [Background] Verschoor MA, Lemmers M, Wekker MZ, Huirne JA, Goddijn M, Mol BW, Ankum WM. Practice variation in the management of first trimester miscarriage in the Netherlands: a nationwide survey. Obstet Gynecol Int. 2014;2014:387860. doi: 10.1155/2014/387860. Epub 2014 Nov 4. PMID 25538770
- [Derived] Hamel CC, Vart P, Vandenbussche FPHA, Braat DDM, Snijders MPLM, Coppus SFPJ. Predicting the likelihood of successful medical treatment of early pregnancy loss: development and internal validation of a clinical prediction model. Hum Reprod. 2022 May 3;37(5):936-946. doi: 10.1093/humrep/deac048. PMID 35333346
- [Derived] Hamel C, Coppus S, van den Berg J, Hink E, van Seeters J, van Kesteren P, Merien A, Torrenga B, van de Laar R, Terwisscha van Scheltinga J, Gaugler-Senden I, Graziosi P, van Rumste M, Nelissen E, Vandenbussche F, Snijders M. Mifepristone followed by misoprostol compared with placebo followed by misoprostol as medical treatment for early pregnancy loss (the Triple M trial): A double-blind placebo-controlled randomised trial. EClinicalMedicine. 2021 Jan 6;32:100716. doi: 10.1016/j.eclinm.2020.100716. eCollection 2021 Feb. PMID 33681738
- [Derived] van den Berg J, Hamel CC, Snijders MP, Coppus SF, Vandenbussche FP. Mifepristone and misoprostol versus misoprostol alone for uterine evacuation after early pregnancy failure: study protocol for a randomized double blinded placebo-controlled comparison (Triple M Trial). BMC Pregnancy Childbirth. 2019 Nov 27;19(1):443. doi: 10.1186/s12884-019-2497-y. PMID 31775677
- See also: The management of early pregnancy loss. Royal College of Obstetricians and Gynaecologists, Green-top Guideline No. 25. — https://www.rcog.org.uk/
- See also: Zwangerschapsafbreking tot 24 weken. Richtlijn Nederlandse Vereniging voor Obstetrie & Gynaecologie. — http://www.nvog.nl
- See also: Cytotec UK SPC (Summary of Product Characteristics). — http://www.medicines.org.uk/emc/medicine/9352
- See also: Mifegyne 200 mg tablets: Summary of Product Characteristics (SmPC) — http://www.exelgyn.com
- See also: Mifepristone - Mifegyne — http://www.farmacotherapeutischkompas.nl
- See also: Erytrocytenimmunisatie en zwangerschap. Versie 2.1, 2009. — http://nvog-documenten.nl/

DOCUMENTS (2):
  • Study Protocol (2019-09-20): https://cdn.clinicaltrials.gov/large-docs/52/NCT03212352/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-03): https://cdn.clinicaltrials.gov/large-docs/52/NCT03212352/SAP_001.pdf